CLINICAL TRIAL: NCT06088394
Title: Effect of Pelvic Floor Exercises Versus Pelvic Floor Exercises and Acupuncture on Overactive Bladder
Brief Title: Effect of Acupuncture Augmented With Pelvic Floor Exercises on Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Ahmed Elsayed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004593
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Overactive Bladder Syndrome
Keywords: pelvic floor exercises and acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: pelvic floor exercises and acupuncture
Who Masked: Participant
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The patients will do pelvic floor exercises and acupuncture (Experimental): The patients will perform pelvic floor exercises and acupuncture 3 times per week for 12 weeks
  Interventions: Device: Acupuncture; Other: pelvic floor exercises
- The patient will do pelvic floor exercises (Experimental): The patient will perform pelvic floor exercises 3 times per week for 12 weeks. pelvic floor muscles exercises involves repetitive contraction and relaxation of the pelvic floor muscles in an attempt to strengthen the muscles .
  Each training session involved three training rounds and each round lasted for five minutes. Women will be instructed to perform PFMC and rest with 10min break between each round. They will be instructed to perform two to three sets of PFE repetitions per day, with 8-10 PFMC lasting for 10 s each set. All women will be asked to document their practice of PFE in PFE diary to assess their compliance.
  Interventions: Other: pelvic floor exercises

INTERVENTIONS:
Device: Acupuncture — Participants will be asked to assume supine lying position on the plinth and the following points will be located then needles will be inserted:
  * CV3,4 &5-40 mm needles at a depth of 1 cun perpendicular insertion.
  * ST 25 bilaterally-40 mm needles at a depth of 1 cun oblique insertion.
  * SP6 & 9, K13&7 bilaterally-25 mm needles at a depth of 0.5 cun perpendicular insertion. A total of 13 needles will be inserted at each session.
  Arms: The patients will do pelvic floor exercises and acupuncture
Other: pelvic floor exercises — pelvic floor muscle exercises can help strengthen pelvic floor muscle, which provides better control of urinary urgency by interfering with urethral-detrusor reflexes and inhibiting detrusor contractions

SUMMARY:
The aim of this study is to investigate the effect of pelvic floor exercises augmented with acupuncture on overactive bladder

DETAILED DESCRIPTION:
Overactive bladder syndrome (OAB) is a common complaint affecting 11.8% of the population. OAB is defined by the International Continence Society as "urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of urinary tract infection or other obvious pathology."Urinary frequency accompanies OAB in 20%-25% of cases, and nocturia is present in 70%-75% of cases. Around one in three people with OAB also experience urinary incontinence. . OAB can be further categorized into "OAB-dry" (urinary incontinence is absent) and "OAB-wet" (urinary incontinence is present). 2 OAB is a long-term condition that reduces quality of life, leading to anxiety and depression and a negative effect on self-esteem.

Pelvic floor exercises and acupuncture play an important role in overactive bladder.This trial has 2 groupes ,one will recieve pelvic floor exercises augmented with acupuncture ,the second will recive pelvic floor exercises only for 12weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients with a clinical diagnosis of idiopathic OAB syndrome. Willingness to take part in the study protocol. Ability to complete outcome measures. Ability to give informed consent. Acupuncture not contra-indicated. Age:50-60 years. Vaginal delivery.

-Parity:2-3times. Body mass index <35kg/m2.

Exclusion Criteria:

* - Evidence of other pathology that may be contributing to OAB symptoms i.e., urinary tract infection or a neurological condition.
* Smoking.
* Taking sedative and hypnotic drugs.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-13 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Oxford scale | 12 weeks
  The scale ranges from 0 to 5 ranging from "no contraction" to "maximal contraction which is assessed by digital palpation using 1 to 2 fingers inserted into the vagina or rectum . This method is reliable to assess improvements in overall function and voluntary control of the PFM necessary for proper voiding

SECONDARY OUTCOMES:
patient perception of intensity and urgency scale (PPIUS) | 12 WEEKS
  A 5-point scale designed for measurement of both urinary urgency and urge incontinence. It has been incorporated into a micturition diary and has been used in OAB clinical trials

OTHER OUTCOMES:
8 Items overative bladder questionnaire | 12 weeks
  : The OAB-V8 asks how bothered one is by the 4 hallmark symptoms of OAB: urinary frequency, urgency, nocturia, and urge incontinence Patients respond on a 6-point Likert scale ranging from 0 (not at all) to 5 (a very great deal), with a maximum possible score of 40. After completing the awareness tool, patients were asked to calculate their scores by adding their responses .
3days bladder diary test | 12 weeks
  It consists of three sheets to be completed by the patient (one for each day) and one evaluation sheet to be completed by the clinician based on the interpretation of the three patient-completed sheets. The patient should record, on the daily sheet, the time they wake up and go to bed and the time and volume of every micturition.

CONTACTS AND LOCATIONS:
Overall Officials: cairo U Egypt, Study Chair — faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes